CLINICAL TRIAL: NCT01729286
Title: A Multi-Center, Prospective, Randomized Study With PriMatrix Dermal Repair Scaffold Moist Wound Therapy and Standard of Care Moist Wound Therapy for the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: Health Economic Assessment of Lower Extremity Diabetic (HEALED) Ulcers With PriMatrix
Acronym: HEALED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEI-007
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PriMatrix Moist Wound Therapy (Active Comparator): sharp debridement, Primatrix, a dressing regimen that maintains a moist wound healing environment, and offloading
  Interventions: Device: PriMatrix Moist Wound Therapy; Other: Standard of Care Moist Wound Therapy
- Standard of Care Moist Wound Therapy (Other): sharp debridement, a dressing regimen that maintains a moist wound healing environment, and offloading
  Interventions: Other: Standard of Care Moist Wound Therapy

INTERVENTIONS:
Device: PriMatrix Moist Wound Therapy — sharp debridement, PriMatrix, a dressing regimen that maintains a moist wound healing environment, and offloading
  Other Names: PriMatrix Dermal Repair Scaffold
  Arms: PriMatrix Moist Wound Therapy
Other: Standard of Care Moist Wound Therapy — sharp debridement, a dressing regimen that maintains a moist wound healing environment, and offloading

SUMMARY:
The objective of this study is to compare the effectiveness of PriMatrix Moist Wound Therapy (MWT) with Standard of Care MWT for the treatment of chronic diabetic foot ulcers in subjects with diabetes mellitus and without significantly compromised arterial circulation.

DETAILED DESCRIPTION:
This study will be a multi-center, prospective, randomized single-blinded study evaluating the efficacy of PriMatrix MWT versus Standard of Care MWT in achieving complete wound closure of chronic diabetic foot ulcers by 12 weeks (84 days). To measure wound recidivism and changes in functional quality of life, each subject will complete the Cardiff Wound Impact Schedule and the SF-36v2™ at three time points during the study i) at initial screening, ii) at completion of treatment phase, and iii)at 24 weeks (post-randomization). Additionally, the data obtained from the SF-36v2™ will be used in an economic evaluation of the treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Type I or Type II diabetes
* A diabetic foot ulcer located on the foot or ankle at least one square centimeter

Exclusion Criteria:

* Suspected or confirmed signs/symptoms of wound infection
* Hypersensitivity to bovine collagen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Complete wound closure | by 12 weeks

SECONDARY OUTCOMES:
Change in predicted medical expenditures between PriMatrix and Standard of Care | over 24 weeks
Change in quality of life measurements between PriMatrix and Standard of Care | between baseline and 24 weeks
Nonserious and serious adverse events | over 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Starinski, DPM, Study Chair — TEI
Locations (18):
- United States (15):
  - University of Southern California, Los Angeles, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Advanced Research Institute of Miami, Miami, Florida
  - Advanced Foot & Ankle Specialists, Tampa, Florida
  - Joseph M. Still Research Foundation, Augusta, Georgia
  - American Health Network, Carmel, Indiana
  - Foot & Andle Center of Mooresville, Mooresville, Indiana
  - Imperial Health, Lake Charles, Louisiana
  - Kansas City Vascular, North Kansas City, Missouri
  - St. Anthony's Medical Center, St Louis, Missouri
  - North Shore Long Island Jewish Comprehensive Wound Healing Center, Lake Success, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Fairfield Medical Center, Lancaster, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
- Puerto Rico (3):
  - Centro Podiatrico del Norte, Arecibo
  - Renier Gonzalez-Cruz, Juana Díaz
  - VA Carribean Healthcare System, San Juan

IPD SHARING:
Plan to Share IPD: No